CLINICAL TRIAL: NCT01018693
Title: Randomized, Double-blind, Placebo-controlled Trial to Determine the Capacity of VAK694 to Elicit Long Term Immune Tolerance When Combined With Subcutaneous Allergen Immunotherapy for the Treatment of Seasonal Allergic Rhinitis
Brief Title: A Study to Determine the Capacity of VAK694 When Combined With Allergen Immunotherapy to Bring About Specific Immune Tolerance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVAK694A2205
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Seasonal allergic rhinitis,; late phase response,; alutard avanz,; immunotherapy,; visual analogue scale,; mini rhinitis quality of life,; immune modulation
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- VAK694 AND Immunotherapy (alutard) (Experimental)
  Interventions: Drug: VAK694; Alutard Avanz SQ
- : VAK694 placebo AND Immunotherapy (alutard) (Experimental)
  Interventions: Drug: VAK694 placebo infusion; Alutard Avanz SQ
- VAK694 placebo AND Immunotherapy (alutard) placebo (Experimental)
  Interventions: Drug: VAK694 placebo infusion; Saline

INTERVENTIONS:
Drug: VAK694; Alutard Avanz SQ
  Arms: VAK694 AND Immunotherapy (alutard)
Drug: VAK694 placebo infusion; Alutard Avanz SQ
  Arms: : VAK694 placebo AND Immunotherapy (alutard)
Drug: VAK694 placebo infusion; Saline
  Arms: VAK694 placebo AND Immunotherapy (alutard) placebo

SUMMARY:
The purpose of the study is to determine whether VAK694 when combined with subcutaneous immunotherapy leads to long term immune tolerance to allergen in individuals with seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* History of atopy, defined as a history of seasonal allergic rhinitis for at least 2 years (in relation to the grass pollen allergy season), and evidence of atopy, defined as a positive skin prick test (wheal difference allergen - negative control at least 3 mm) to grass pollen allergen at screening.
* Male or female subjects aged between 18 and 60 years (inclusive)
* Female subjects must be of non-childbearing potential
* Subjects must weigh at least 50 kg with a body mass index (BMI) within the range of 18 to 32 kg/m2 (inclusive)
* Informed consent

Exclusion Criteria:

* Treatment with intranasal corticosteroids within 28 days prior to the first dose.
* History of asthma with treatment with inhaled or systemic corticosteroids within 6 months of the first dose.
* History of COPD.
* Any exposure to human monoclonal or polyclonal antibodies.
* Any allergy immunotherapy within 3 years prior to screening.
* Any prior grass pollen allergy immunotherapy.
* FEV1 < 70% of predicted at screening or baseline.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Intra-dermal late phase response to allergen Measure: Wheal diameter | 10-12 months

SECONDARY OUTCOMES:
To evaluate the immunomodulatory activity of VAK694 Measure: IgE/IgG, Th1/Th2 cytokine expression, Treg induction | 10-12 months
To assess the effects of VAK694 combined with SCIT on the symptoms of seasonal allergic rhinitis Measure: mini-Respiratory Quality of Life Questionnaire (RQLQm) and visual analogue scale (VAS) | 10-12 months
To preliminarily assess the ability of VAK694 to reduce the side-effects of subcutaneous immunotherapy Measure: Frequency and severity of local and systemic reactions to immunotherapy | 10-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigator Site, London, United Kingdom

REFERENCES:
- See also: Related Info — http://www.hayfeverlondon.net